CLINICAL TRIAL: NCT06221111
Title: Rimegepant, a CGRP Antagonist, in the Treatment of Visceral Sensation and Chronic Abdominal Pain: A Pilot Study
Brief Title: Comparison of Rimegepant and Placebo for Pain in IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Professor of Medicine, Pharmacology and Physiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-006559
Record Dates: First submitted 2024-01-05; First posted 2024-01-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: pain, IBS, CGRP, rimegepant, antagonist
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain; Ichthyosis Bullosa of Siemens | interventions — rimegepant sulfate

STUDY DESIGN:
Intervention Model Description: randomized, double-blind placebo-controlled trial of rimegepant at doses and route of administration approved by the FDA for the prophylaxis of migraine headache.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: concealed allocation; blinded provision of assigned medication through research pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- rimegepant (Experimental): * Rimegepant 75mg oral dissolving tablet (ODT)
  * Formulation and Dosing as FDA-approved for Migraine Prevention: 75 mg Every Other Day (EOD) for 4 weeks/30 days
  Interventions: Drug: Rimegepant 75 MG [Nurtec]
- placebo (Placebo Comparator): Placebo ODT appearing identical to the experimental formulation and administered every other day for 4 weeks/30 days
  Interventions: Drug: Rimegepant 75 MG [Nurtec]

INTERVENTIONS:
Drug: Rimegepant 75 MG [Nurtec] — placebo controlled trial
  Other Names: placebo

SUMMARY:
The primary aim of this study is to evaluate the efficacy of rimegepant on abdominal pain scores in participants with non-constipation IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) and, particularly, the pain component of IBS lack effective treatments. Antispasmodics, antidepressants and hypnotherapy have all been proposed for the treatment of pain. Their effectiveness in clinical practice is disappointing, despite meta-analyses suggesting efficacy. The study hypotheses are: that rimegepant will be safe, well-tolerated, and will improve abdominal pain in participants with non-constipation IBS. The primary aim is to evaluate the efficacy of rimegepant on abdominal pain scores in participants with non-constipation IBS. Secondary aims of this study are:

* 1: To describe the effect of rimegepant on rectal compliance in participants with IBS and chronic abdominal pain.
* 2: To evaluate the effects of rimegepant on rectal sensation based on ascending method of limits and on graded rapid phasic distensions in participants with non-constipation IBS and chronic abdominal pain.
* 3: To evaluate effects of rimegepant on overall colonic transit in participants with non-constipation IBS and chronic abdominal pain.
* 4: To evaluate safety of rimegepant in participants with non-constipation IBS and chronic abdominal pain Methods: IBS-pain participants will be selected according to the Rome III criteria. Trial participants will continue to receive the same medical therapy throughout the baseline and treatment periods. The study design is a randomized, double-blind placebo-controlled trial of rimegepant at doses and route of administration approved by the FDA for the prophylaxis of migraine headache.

The trial period will consist of a two week run-in period, and 4 week treatment period. Participants will complete a daily diary regarding abdominal pain and stool consistency. They will also complete questionnaires studies of anxiety and depression and IBS-QOL.

An established and validated method using rectal barostat device will be used to measure rectal compliance and sensation. The standard scintigraphic method to measure colonic transit established in the Clinical Research Trials Unit (CRTU) at Mayo Clinic Rochester will be used to evaluate changes in colonic transit.

Anticipated results and Significance: Rimegepant, at doses and mode of administration approved by FDA for the prophylaxis of migraine headache, will be efficacious in the reduction of abdominal pain and rectal sensation in participants with non-constipation IBS and abdominal pain.

This study will provide an early signal of efficacy that may lead to future randomized, controlled trials.

ELIGIBILITY:
Twenty-four participants with non-constipation IBS and chronic abdominal pain will be recruited for enrollment. Participants will meet specific Rome III IBS diagnostic criteria.

Inclusion criteria:

* Participants will be 18-70 years of age.
* Participants will have non-constipation IBS [that is IBS-D (diarrhea), IBS-M (mixed), or IBS-U (unspecified)] with chronic abdominal pain diagnosed in their medical records at Mayo Clinic with chronic pain documented for ≥ 3 months.
* Participants will have subjective pain ratings of ≥ 30 on the 100 mm VAS during at least 1 of the 2 run-in weeks for enrollment.
* Participants will be capable of providing informed consent.

Exclusion criteria:

* Diagnosis of moderate-severe depression as per BDI ≥18;
* Alcohol or illicit substance dependence or abuse in the past 12 months;
* Dementia, unprovoked seizure history, seizure disorder;
* Pregnancy (all women of childbearing potential will be required to have a negative pregnancy test prior to initiation, and will be on a highly effective method of contraception, as detailed in the consent form);
* Significant change or increase in antidepressant or pain medications within the last four weeks; significant change in primary treatment interventions for pain in the past four weeks;
* Medically unstable
* Severe hepatic or renal impairment, such as baseline AST or ALT ≥ 2.5 X upper normal limit or end-stage renal disease with estimated glomerular filtration rate or creatinine clearance <15mL/min. Although Rimegepant is rarely associated with abnormal circulating liver enzymes, we shall exclude patients with baseline AST or ALT equal to or greater than 2.5 times the upper limit of normal.
* Concomitant use of strong CYP3A4 inhibitors and strong or moderate CYP3A4 inducers.
* Participants who report nausea several times per week or daily on the baseline bowel disease questionnaire (question # 16) will be excluded from the study because of the low risk of nausea induced by the treatment which was estimated at approximately 3% for rimegepant compared to 1% for placebo.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
abdominal pain | daily over 4 weeks
  daily abdominal pain scores measured on 100mm Visual analog scale in participants with non-constipation IBS with 0 and 100 as minimum and maximum values and higher scores indicating worse pain .

SECONDARY OUTCOMES:
rectal sensation | on final day of 4 week study
  rectal sensation based on ascending method of limits and on graded phasic distensions
rectal compliance | on final day of 4 week study
  rectal compliance in participants with non-constipation IBS and chronic abdominal pain
colonic transit | during days 26-28 of 4 week study
  overall colonic transit by scintigraphy
safety based on adverse effects | during the 4 week study
  evaluate safety of rimegepant in non-constipation IBS and chronic abdominal pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No